CLINICAL TRIAL: NCT00588367
Title: CT Perfusion of Pancreatic Cancer and Chronic Pancreatitis: Feasibility Study
Brief Title: CT Pancreas Perfusion
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Naoki Takahashi, Principal Investigator, Mayo Clinic
Other Study IDs: 360-06
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Chronic Pancreatitis; Autoimmune Pancreatitis
Keywords: Inflammation; Pancreas; Chronic pancreatitis; Alcoholic pancreatitis; Carcinoma, pancreatic ductal; Pancreatic neoplasms
MeSH Terms: conditions — Pancreatitis, Chronic; Autoimmune Pancreatitis; Inflammation; Pancreatitis, Alcoholic; Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Suspected pancreatic ductal adenocarcinoma.
  Interventions: Device: Mayo Interactive Breath Hold Monitor
- 2: Chronic pancreatitis and slated for decompression treatment.
  Interventions: Device: Mayo Interactive Breath Hold Monitor
- 3: Autoimmune pancreatitis.
  Interventions: Device: Mayo Interactive Breath Hold Monitor

INTERVENTIONS:
Device: Mayo Interactive Breath Hold Monitor — Biofeedback device

SUMMARY:
1. Pancreatic CT perfusion with a biofeedback breathing belt worn by the participant, and using novel post-processing techniques, is a reliable method which can be used to differentiate between pancreatic cancer, chronic pancreatitis, and autoimmune pancreatitis.
2. Pancreatic CT perfusion can be used to monitor patients undergoing decompression treatment (endoscopic retrograde cholangiopancreatography with stent placement) for painful chronic pancreatitis, and the change in the pancreatic perfusion parameters correlate with the change in the pain parameters (pain scale and analgesic use).
3. Pancreatic CT perfusion parameters can be calculated using surrogate scan data sets at specific time points to replace the continuous scanning.

ELIGIBILITY:
Inclusion Criteria:

1. a. Suspected pancreatic adenocarcinoma, age 35 to 99 years.
2. a. Chronic pancreatitis with chronic pain, age 18 to 99 years. Must be a confirmed diagnosis by either CT, endoscopic ultrasound (EUS), or endoscopic retrograde cholangiopancreatography (ERCP).

2b. To undergo endoscopic or surgical decompression with 0 to 10 days of first study visit CT perfusion scan.

2c. To answer pain questionnaire before first CT perfusion scan.

2d. To return within three weeks to three months after decompression treatment for another CT perfusion scan and complete the second pain questionnaire.

3a. Autoimmune pancreatitis, age 18 to 99 years either with diffuse or focal swelling of the pancreas confirmed by CT, MRI, or EUS or

3b. Irregular narrowing of the pancreatic duct on ERCP and either elevated serum immunoglobulin G4 (IgG4), or histological confirmation.

Exclusion Criteria:

1a. Pancreatic ductal adenocarcinoma tumors with vascular involvement but without vascular occlusion.

1. b. Pancreatic ductal adenocarcinoma tumors less than 2 cm in size.
2. a. Chronic pancreatitis with diffuse and extensive pancreatic calcification.
3. a. Autoimmune pancreatitis with a prior pancreas surgery or steroid treatment for autoimmune pancreatitis .

Any Cohort:

4. Pregnant.

5. Prior iodine contrast reactions.

6. Iodine allergy.

7. Decreased kidney function being a serum creatinine greater than 1.5mg/dl.

8. Any contraindication to having a CT scan with iodine contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic patients being seen in Pancreas Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
A reproducible technique to measure CT perfusion parameters may provide a method for non-invasively monitoring tumor response during treatment, or differentiating between autoimmune and chronic pancreatitis. | Three weeks to three months for chronic pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Takahashi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States